CLINICAL TRIAL: NCT06782321
Title: Centering Emotional Recovery Post-Stroke
Brief Title: Emotional Recovery Post-Stroke
Acronym: eWELL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: The Duke Endowment (Other)
Responsible Party: Principal Investigator, Michelle Woodbury, Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00138136
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Stroke; Mental Health Wellness 1
Keywords: Rehabilitation Studies; Stroke; Stroke Recovery
MeSH Terms: conditions — Stroke | interventions — Speech Therapy

STUDY DESIGN:
Intervention Model Description: Randomized rehabilitation clinical trial with adaptive design. At study midpoint, a preliminary analysis will identify the intervention showing the greatest effect on the majority of the primary outcome measures. Subsequently, the randomization ratio will be adapted to 2:1 in favor of that intervention
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- modified Cognitive Behavioral Therapy + Telerehabilitation Occupational or Speech Therapy (Experimental)
  Interventions: Behavioral: modified Cognitive Behavioral Therapy (mCBT); Behavioral: Occupational or Speech Therapy
- Telerehabilitation Occupational or Speech Therapy (Active Comparator)
  Interventions: Behavioral: Occupational or Speech Therapy

INTERVENTIONS:
Behavioral: modified Cognitive Behavioral Therapy (mCBT) — The theoretical model underling Cognitive Behavioral Therapy (CBT) explains the interaction of thoughts, feelings, and behaviors during life situations. This model suggests that a person's thoughts/feeling/behaviors affect their functioning during life situations. This contrasts with a common belief that one's functioning during life situations is the only way to effect thoughts/feelings/behaviors. Applied to stroke, this model suggests that the stroke survivor can alter his/her functioning during life situations by altering his/her thoughts/feelings/behaviors. The purpose of CBT is to empower the person with the skills to alter his/her thoughts/feelings/behaviors in order to positively affect function in life situations.
  The mCBT intervention includes 4 elements: psychoeducation, education about unhelpful thinking, behavioral activation therapy, education on sleep hygiene, and relaxation training.
  Arms: modified Cognitive Behavioral Therapy + Telerehabilitation Occupational or Speech Therapy
Behavioral: Occupational or Speech Therapy — If the participant demonstrates aphasia of any severity level on the Revised Western Aphasia Battery (WAB-R) assessment given at the PRE session, the subject will receive ST, provided by a Speech Language Pathologists (SLP), stroke telerehabilitation. If there is no aphasia, the subject will receive OT stroke telerehabilitation.
  The OT and ST stroke telerehabilitation sessions will utilize a similar metacognitive strategy training approach which is focused on enabling the stroke survivor to re-engage with meaningful life activities. In the Occupational Therapy literature this approach is called Cognitive Orientation to Occupational Performance (CO-OP) and in the Speech Language Pathology Literature this approach is called the Life Participation Approach to Aphasia (LPAA).
  Telerehabilitation CO-OP and LPAA within the OT or ST session include three common elements: Shared decision-making for goal setting, guidance/coaching from the therapist, and self-evaluation.

SUMMARY:
The purpose of this study is to evaluate whether adding an emotional wellness component to occupational therapy (OT) and/or speech therapy (ST) telerehabilitation improves overall emotional well-being and activity participation for people with stroke.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate whether adding an emotional wellness component to occupational therapy (OT) and/or speech therapy (ST) telerehabilitation improves overall emotional well-being and activity participation for people with stroke. Participants will complete 9 telerehabilitation therapy sessions over 8 weeks. These sessions will take place over a video visit using a personal device (phone, tablet, or computer). Each session will last about 1 hour. Sessions will focus on occupational therapy and/or speech therapy depending on the participant's stroke-related movement and/or language deficits. Each study participant will be randomly assigned to one of two intervention groups. Both groups will include OT or ST; however, one group will include an emotional wellness component using a modified version of Cognitive Behavioral Therapy. Participants will also complete 2 assessment visits, one before the telerehabilitation begins and one after the telerehabilitation program ends. The assessment visits will also take place via a video visit using a personal device. Assessments include measures of emotional well-being, quality of life, activity engagement, arm/hand movement, communication/language skills, balance, and ability to perform daily activities.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported stroke-related deficits in emotional wellness such as anxiety, sleep disturbance, dread, fear, loss of hope, sadness.
* Have experienced ischemic or hemorrhagic stroke at least 30 days prior
* Stroke-related aphasia and/or upper extremity hemiparesis
* Aged 21 years or older
* English as primary language
* Have corrected vision to be able to read text on a screen
* Able to participate fully in the study's tele-rehabilitation (Aim 1) and/or virtual group programing (Aim 2) with personally owned device (i.e., phone, tablet, or laptop) and personal Wi-Fi connection or cellular service
* Cognitive, language, and motor capacity to participate fully in the study's assessment session as per the judgment of the licensed, experienced stroke tele-rehabilitation occupational or speech therapist

Exclusion Criteria:

* Unable to follow 1-2 step instructions given by the study team member during the informed consent procedures.
* Pain that interferes with ability to participate in the study's upper extremity movement tasks.
* Have impaired decision making capacity as determined by the U-ARE protocol for assessing capacity to provide informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Warwick-Edinburgh Mental Wellbeing Scale (WEMWS) | Baseline, pre-intervention and immediately after the intervention, Week 8.
  14-item scale of mental well-being rated by participants on a 5-point scale (1=low, 5=high). Summed item ratings are reported out of 70 points so that higher scores indicate greater mental wellbeing.
Patient Specific Functional Scale (PSFS) | Baseline, pre-intervention and immediately after the intervention, Week 8.
  A patient-reported measure of task-goal identification and difficulty performing the task on a 0-10-point ordinal scale with higher ratings indicating greater satisfaction with task performance.
Stroke and Aphasia Quality of Life Scale (SAQoL) | Baseline, pre-intervention and immediately after the intervention, Week 8.
  39-item stroke-specific measure of health-related quality of life rated by participants on a 5-point scale (1 = couldn't do it at all, 5 = no trouble at all). An overall mean score is computed as well as three domain scores: physical, communication, and psychosocial. Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Woodbury, PhD, Principal Investigator — Medical University of South Carolina; Lisa McTeague, PhD, Principal Investigator — Medical University of South Carolina; Deena Blackett, PhD, Principal Investigator — University of Central Florida
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ayerbe L, Ayis SA, Crichton S, Wolfe CD, Rudd AG. Natural history, predictors and associated outcomes of anxiety up to 10 years after stroke: the South London Stroke Register. Age Ageing. 2014 Jul;43(4):542-7. doi: 10.1093/ageing/aft208. Epub 2013 Dec 26. PMID 24375225
- [Background] Hackett ML, Pickles K. Part I: frequency of depression after stroke: an updated systematic review and meta-analysis of observational studies. Int J Stroke. 2014 Dec;9(8):1017-25. doi: 10.1111/ijs.12357. Epub 2014 Aug 12. PMID 25117911
- [Background] Bhattacharjee S, Axon DR, Goldstone L, Lee JK. Patterns and Predictors of Depression Treatment among Stroke Survivors with Depression in Ambulatory Settings in the United States. J Stroke Cerebrovasc Dis. 2018 Mar;27(3):563-567. doi: 10.1016/j.jstrokecerebrovasdis.2017.09.047. Epub 2017 Oct 31. PMID 29097059
- [Background] Harrison RA. A simple pattern for Plastazote boots. Physiotherapy. 1984 Mar;70(3):114-5. No abstract available. PMID 6718567
- [Background] Kowalska K, Krzywoszanski L, Dros J, Pasinska P, Wilk A, Klimkowicz-Mrowiec A. Early Depression Independently of Other Neuropsychiatric Conditions, Influences Disability and Mortality after Stroke (Research Study-Part of PROPOLIS Study). Biomedicines. 2020 Nov 17;8(11):509. doi: 10.3390/biomedicines8110509. PMID 33213019
- [Background] McKevitt C, Fudge N, Redfern J, Sheldenkar A, Crichton S, Rudd AR, Forster A, Young J, Nazareth I, Silver LE, Rothwell PM, Wolfe CD. Self-reported long-term needs after stroke. Stroke. 2011 May;42(5):1398-403. doi: 10.1161/STROKEAHA.110.598839. Epub 2011 Mar 24. PMID 21441153
- [Background] Skolarus LE, Lisabeth LD, Burke JF, Levine DA, Morgenstern LB, Williams LS, Pfeiffer PN, Brown DL. Racial and Ethnic Differences in Mental Distress among Stroke Survivors. Ethn Dis. 2015 Spring;25(2):138-44. PMID 26118139
- [Background] HRSA. Behavioral Health Workforce, 2023. In: HRSA, editor.: National Center for Health Workforce Analysis; 2023.
- [Background] Services UDoHaH. South Carolina Mental Health Health Professional Shortage Areas (HPSA): GIS Office of Information Technology; 2023 [updated 03-07-2023]. Available from: https://scdhec.gov/sites/default/files/media/document/HPSA-Mental-Health-2023.pdf.
- [Background] Hamilton RKB, Phelan CH, Chin NA, Wyman MF, Lambrou N, Cobb N, Kind AJH, Blazel H, Asthana S, Gleason CE. The U-ARE Protocol: A Pragmatic Approach to Decisional Capacity Assessment for Clinical Research. J Alzheimers Dis. 2020;73(2):431-442. doi: 10.3233/JAD-190457. PMID 31868663
- [Background] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300